CLINICAL TRIAL: NCT03449342
Title: Safety of Turoctocog Alfa for Prophylaxis and Treatment of Bleeding Episodes in Previously Treated Patients With Moderate or Severe Haemophilia A in India
Brief Title: Research Study to Look at Side Effects During Regular Injection With Factor VIII Medicine Named Turoctocog Alfa for a 8 Weeks Period
Acronym: guardian 10
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-4304; 2017-002281-46 (Registry Identifier: EudraCT); U1111-1179-5950 (Other: World Health organization (WHO))
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Turoctocog alfa (Experimental): Previously treated moderate or severe haemophilia A patients will receive routine prophylaxis treatment and treatment of bleeding episodes.
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Patients will receive standard prophylaxis treatment and treatment of bleeding episodes, according to label. Trial product will be administered as intravenous injections (i.v.)

SUMMARY:
This study will test the well-known medicine turoctocog alfa for any side effects. The purpose is to test turoctocog alfa for any side effects in the Indian population. The participants will get turoctocog alfa. Turoctocog alfa is already a well-known medicine in India, and can be prescribed by the study doctor. The participants will get an injection every second day or 3 times per week. This is decided by the study doctor. The study doctor will decide the amount and how often the participants must take the medicine. The study will last for about 16 weeks. The participants will have 5 visits with the study doctor. If the participants agree to participate in this study, the participants will receive the first injection at the second visit, thereafter the participants will be trained to do the injection by themself.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Male, age above or equal to 12 years at the time of signing informed consent - Patients with the diagnosis of congenital moderate or severe Haemophilia A based on medical records. (FVIII below or equal to 5%) - Documented history of at least 150 EDs (exposure days) to FVIII containing products Exclusion Criteria: - Confirmed inhibitors to FVIII (above or equal to 0.6 BU) at screening as assessed by central laboratory - History of FVIII inhibitors - Known or suspected hypersensitivity to trial product(s) or related products - Previous participation in this trial. Participation is defined as signed informed consent - Participation in any clinical trial of an approved or non-approved investigational medicinal product within 1 month before screening (visit 1) - Any disorder, except for conditions associated with haemophilia A, which in the investigator's opinion might jeopardise patient's safety or compliance with the protocol - Immunocompromised patients due to HIV infection (defined as viral load above or equal to 400.000 copies/mL and/or CD4+ lymphocyte count below or equal to 200/μL). HIV status and CD4+ lymphocyte count /viral load results may be obtained at screening or from available medical records; results must be not older than 6 months - Known congenital or acquired coagulation disorders other than haemophilia A - Mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Ludhiana, Punjab
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 10 sites in India.
Groups:
- Adolescents (12 - <18 Years); Adults (≥18 Years): Participants were to receive prophylactic (preventive) treatment of turoctocog alfa as intravenous (i.v.) injections at a frequency of 'every second day' or '3 times a week' at a dose in the range of 20-50 IU/kg at the investigator's discretion. Dosing for prophylaxis was according to the approved prescribing information. The total treatment duration for each participant was 8 weeks. Bleeds were treated with one or more turoctocog alfa intravenous (i.v.) bolus injections. The individual dose levels were decided by the investigator based on recommendations from the World Federation of Hemophilia (WFH). Participants who underwent surgery were treated with turoctocog alfa according to WFH recommendations.
Period: Overall Study
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Started | 10 | 50
Completed | 10 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years) | Total
Number analyzed (Participants) | 10 | 50 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.90 (1.91) | 27.10 (7.28) | 24.90 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 50 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 50 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 50 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Confirmed FVIII Inhibitor Development (≥ 0.6 BU)
Description: The number of participants who confirmed the presence of FVIII inhibitor development (≥ 0.6 BU) during 8 weeks of treatment period.
Time Frame: Weeks 0-8
Population: Results are based on the full analysis set (FAS), that included all dosed participants with data after dosing during 8 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 10 | 50
Participants | 0 | 0

2. Secondary Outcome: Incidence of Adverse Drug Reactions (ARs) and Serious Adverse Reactions (SARs)
Description: Incidence of adverse drug reactions (ARs) and serious adverse reactions (SARs) were calculated as the number of adverse reactions per patient years. All presented ARs and SARs are treatment emergent and related to trial product, which were defined as the events reported after trial product administration until the follow-up, 12 weeks after first treatment.
Time Frame: Weeks 0-12
Population: Results are based on the safety analysis set (SAS), that included all dosed participants with data after dosing during 8 weeks of treatment.
Measure: Number; unit: Number of ARs per patient years
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 10 | 50
Number of ARs per patient years
  Adverse drug reaction | 0 | 0
  Serious adverse reactions | 0 | 0

3. Secondary Outcome: Number of Bleeding Episodes With Successful Haemostatic Effect of Turoctocog Alfa
Description: The haemostatic effect (HE) of turoctocog alfa when used for treatment of bleeding episodes was evaluated during 8 weeks of treatment. Successful haemostatic effect means the haemostatic response when used for treatment of a bleeding episode was either excellent or good. Excellent haemostatic respose: Abrupt pain relief and/or clear improvement in objective signs of bleeding episode within approximately 8 hours after a single injection. Good haemostatic response: Definite pain relief and/or improvement in signs of bleeding episode within approximately 8 hours after an injection, but possibly requiring more than 1 injection for complete resolution.
Time Frame: Weeks 0-8
Population: Results are based on the FAS that included all dosed participants with data after dosing during 8 weeks of treatment. "Overall Number of Participants Analyzed" = Number of participants with bleeding episodes treated with turoctocog alfa.
Measure: Number; unit: Bleeding episodes with successfull HE
Units Other Than Participants: bleeding episodes
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 2 | 17
Number analyzed (bleeding episodes) | 3 | 46
Bleeding episodes with successfull HE | 2 | 38

4. Secondary Outcome: Total Annualised Consumption of Turoctocog Alfa
Description: Total consumption of turoctocog alfa was evaluated during 8 weeks of treatment and it was presented as IU of turoctocog alfa/kg body weight (BW) per year per participant.
Time Frame: Weeks 0-8
Population: Results are based on the FAS that included all dosed participants with data after dosing during 8 weeks of treatment.
Measure: Mean (Standard Deviation); unit: IU/kg BW/year/participant
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 10 | 50
IU/kg BW/year/participant | 7030 (1053) | 6086 (1735)

5. Secondary Outcome: Incidence of Allergic or Infusion Reactions Related to the Trial Product
Description: Incidence of allergic or infusion reactions related to trial products were calculated as the number of reactions per patient years. Allergic reactions are a class of adverse events related to allergy.
Time Frame: Weeks 0-12
Population: Results are based on the SAS, that included all dosed participants with data after dosing during 8 weeks of treatment.
Measure: Number; unit: Number of reactions per patient years
Arm/Group | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 10 | 50
Number of reactions per patient years | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 - 12 (8 weeks of treatment period + 4 weeks of follow-up period).
Description: All the adverse events are based on the safety analysis set (SAS) which included all dosed participants with data after dosing.
Groups:
- Adults (>=18 Years): Participants were to receive prophylactic (preventive) treatment of turoctocog alfa as intravenous (i.v.) injections at a frequency of 'every second day' or '3 times a week' at a dose in the range of 20-50 IU/kg at the investigator's discretion. Dosing for prophylaxis was according to the approved prescribing information. The total treatment duration for each participant was 8 weeks. Bleeds were treated with one or more turoctocog alfa intravenous (i.v.) bolus injections. The individual dose levels were decided by the investigator based on recommendations from the World Federation of Hemophilia (WFH). Participants who underwent surgery were treated with turoctocog alfa according to WFH recommendations.
Arm/Group | Adolescents (12 - <18 Years) | Adults (>=18 Years)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/50
Other Adverse Events (participants affected / at risk) | 2/10 | 2/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents (12 - <18 Years) (N=10) | Adults (>=18 Years) (N=50)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03449342/Prot_SAP_000.pdf